CLINICAL TRIAL: NCT06602557
Title: " a Randomized Pilot Study of the Benefit of Nebulized Amikacin in the Treatment of Gram-negative Bacillus Pneumonia Acquired During Mechanical Ventilation in Patients Receiving Extracorporeal Membrane Veno-arterial Oxygenation (ECMO-VA). "
Brief Title: " a Randomized Pilot Study of the Benefit of Nebulized Amikacin in the Treatment of Gram-negative Bacillus Pneumonia Acquired During Mechanical Ventilation in Patients Receiving Extracorporeal Membrane Veno-arterial Oxygenation (ECMO-VA)."
Acronym: NAVAP-ECMO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAVAP-ECMO
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: Pneumonia, Bacterial; Extracorporeal Membrane Oxygenation
Keywords: ECMO; Hospital acquired pneumonia; Antibiotic nebulization; Pharmacokinetic
MeSH Terms: conditions — Pneumonia, Bacterial; Healthcare-Associated Pneumonia | interventions — Amikacin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amikacine nebulization associated with Standard of care (Experimental)
  Interventions: Drug: Amikacin
- Standard of care (Active Comparator)
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Amikacin — Patients included in the inhaled amikacin group will receive inhaled antibiotic therapy by nebulization of amikacin at a dose of 25 mg/kg in 1 daily dose (+/- 3 hours apart), within 6 hours of randomization and for a total duration of 5 days.
  Arms: Amikacine nebulization associated with Standard of care
Drug: Standard of care — Patients included in the standard of care group will not receive any nebulization. They will receive Standard care alone.
  Arms: Standard of care

SUMMARY:
Pneumonia are the most frequent infectious complication in patients on Extracorporeal Membrane Oxygenation Veno-arterial (ECMO-VA), with a treatment failure rate of around 40%, even though antibiotic therapy is tailored to the germs identified. One hypothesis to explain this particularly high failure rate is the reduced pulmonary blood flow associated with ECMO offloading of the heart. Although there are no data to date on the pulmonary penetration of antibiotics in patients undergoing VA-ECMO, this phenomenon of pulmonary hypoperfusion could contribute to altering the alveolocapillary diffusion of antibiotics, thereby reducing their concentration in the pulmonary parenchyma.

Our hypothesis is that amikacin nebulization could increase bacterial clearance and, ultimately, limit treatment failure or recurrence of gram-negative bacilli (GNB) pneumonia in patients undergoing VA-ECMO.

ELIGIBILITY:
Inclusion Criteria:

1. Patient 18 years or older
2. Circulatory assistance by veno-arterial ECMO for at least 24 hours prior to documentation of pneumonia
3. Invasive mechanical ventilation
4. Diagnostic suspicion of pneumonia based on evocative criteria (presence of at least 2 of the following criteria): fever (superior to 38. 5°C), hypothermia (inferior to 36.0°C), hyperleukocytosis (superior to 11 × 10^9 l-1) or leukopenia (inferior to 4 × 10^9 l-1), purulent tracheobronchial secretions, altered oxygenation with need to increase FiO2 on ECMO or ventilator for the same SaO2 or PaO2 target, new or persistent pulmonary infiltrate(s) on chest x-ray in bed, or image suggestive of pneumonia on chest CT, or consolidation of appearance suggestive of an infectious origin on pulmonary ultrasound.
5. And microbiological confirmation of Gram-negative ventilator-associated pneumonia by quantitative culture on bronchoalveolar lavage (BAL, significance threshold superior to 10^4 CFU/ml) or protected distal sampling (PDP, significance threshold superior to 10^3 CFU/ml).
6. Probabilistic antibiotic therapy with piperacillin - tazobactam
7. Informed consent obtained from the patient or trusted support person if unable to consent at the time of inclusion, or inclusion procedure in emergency situations.
8. Patient affiliated to social security (excluding AME)

Exclusion Criteria:

1. Known allergy to amikacin or another aminoglycoside or to an auxiliary drug or to any of their excipients.
2. Contraindication to the administration of amikacin or its excipients listed in the summary of product characteristics.
3. Contraindication to the administration of an auxiliary drug or to one of its excipients listed in the summary of product characteristics.
4. Contraindications to nebulization
5. Intravenous antibiotic therapy started more than 72 hours before randomization
6. Probabilistic venous antibiotic therapy other than piperacillin - tazobactam
7. Administration of inhaled antibiotics within 7 days prior to inclusion
8. Positive pregnancy test for women of childbearing potential
9. Presence of HIV infection with CD4 count inferior to 200 cells/mm3 or fungal lung infection or pulmonary abscess or empyema
10. Presence of renal insufficiency with creatinine clearance inferior to 15 ml/min, with the exception of patients receiving continuous renal purification or daily hemodialysis sessions as part of their intensive care unit management.
11. Patent moribund (SAPS II superior to 75) or high probability of death within 48 hours
12. Patient under legal protection (curatorship, guardianship or safeguard of justice)
13. Participating in another interventional clinical trial or within the exclusion period at the end of a previous study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Bacterial eradication rate | Day 5
  Bacterial eradication rate, defined as absence of germs on direct examination and negative culture of a tracheal aspirate taken on day 5 (D5) after randomization and at least 12 hours after the last administration of inhaled amikacin.

SECONDARY OUTCOMES:
Clinical cure rate | Day 5
  Clinical cure rate, defined as disappearance of clinical signs suggestive of pneumonia, biological inflammatory syndrome and correction of haematosis disorders, at D5.
Pneumonia persistence rate | Day 5
  Pneumonia persistence rate defined as the presence of the pathogen identified at a significant level on culture of tracheal aspirate at D5.
Change in clinical pulmonary infection score (CPIS) | Day 0 to Day 5
  Difference between CPIS score at D5 and CPIS score at randomization.
Change in pulmonary aeration score | Day 0 to Day 5
  Difference between ultrasound pulmonary aeration score at D5 and pulmonary aeration score at randomization.
Adverse events | Day 0 to Day 5
  Quantifying and analysing adverse events and serious adverse events
Pharmacokinetic analysis of piperacillin tazobactam | Day 1
  Pharmacokinetic analysis of plasma concentrations of the piperacillin - tazobactam combination
Alveolar fluid penetration ratio of piperacillin-tazobactam | Day 1
  Measurement of the alveolar fluid penetration ratio (AUC* alveolar fluid / AUC plasma) of piperacillin-tazobactam in patients on ECMO-VA after 2 days of intravenous antibiotic administration.
  *Area Under the Curve
Pharmacokinetic analysis of Amikacin | Day 1 to Day 5
  Measurement of the plasma concentration of Amikacin in patients on ECMO-VA in the treatment group between D1 and D5.
Alveolar fluid concentration of Amikacin | Day 1
  Measurement of the alveolar fluid concentration of Amikacin in patients on ECMO-VA after one nebulization in the treatment group (after 24 hours of treatment)

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor.
Access Criteria: Researchers who provide a methodologically sound proposal.